CLINICAL TRIAL: NCT03164291
Title: Clinical Efficacy of Rifabutin in the Treatment of Serious and Life Threatening Infections Due to Mycobacterium Avium Complex, or Drug Resistant Mycobacterium Tuberculosis, or Other Drug Resistant Mycobacterium
Brief Title: Effectiveness of Rifabutin in the Treatment of Mycobacterium Avium Complex
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at Tyler (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Richard J. Wallace, Jr., M.D., Chairman Department of Microbiology, The University of Texas Health Science Center at Tyler
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 072
Record Dates: First submitted 2008-01-14; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Nontuberculous Mycobacterial Infections
Keywords: MAC and NTM
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection | interventions — Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rifabutin (Experimental): Treatment of adults with chronic Mycobacterium avium-intracellulare complex lung infections or other NTM disease who fail therapy with other drugs ( i.e., rifampin)
  Interventions: Drug: Rifabutin

INTERVENTIONS:
Drug: Rifabutin — Rifabutin dosage dependent on clinical factors such as age, weight, and patient-specific health status
  Other Names: mycobutin

SUMMARY:
Treatment of adults with chronic Mycobacterium avium-intracellulare complex lung infections who have failed or are intolerant of rifampin.

Rifabutin may be a reasonable alternative agent in patients who fail rifampin or or intolerant of rifampin.

DETAILED DESCRIPTION:
Rifabutin dosage 150-300 mg daily( depending upon age, and clinical conditions) in NTM patients who fail treatment with rifampin.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and older with positive acid-fast bacilli smears and cultures for drug-resistant mycobacteria

Exclusion Criteria:

* Children less than 18 years of age
* Pregnancy
* Low platelet count, except with very serious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 1984-06; Primary Completion 2006-09 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Clinical and microbiological outcomes (e.g. clinical symptoms, laboratory cultures) | 6 mos
  neg cultures X3( sputum conversion)

SECONDARY OUTCOMES:
Microbiological Cultures | 1year
  neg cultures for 1 yr on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Wallace, Jr, M.D., Principal Investigator — The University of Texas Health Center at Tyler; William B Girard, MD, Study Chair — University of Texas Health Science Center IRB Chair
Locations (1):
- The University of Texas Health Science Center at Tyler, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: No